CLINICAL TRIAL: NCT06884878
Title: Multi-omic Approach to Cancer Diagnosis: the Italian Network of Excellence for Advanced Diagnosis (INNOVA)
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Other Study IDs: INNOVA
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Multi-omic approach to cancer diagnosis. — To assess the impact of intratumoral heterogeneity on the effectiveness of targeted therapies and immunotherapy.

SUMMARY:
The INNOVA project aims to create an advanced multidisciplinary diagnostic platform to support the Italian healthcare system and translational research. In this context, WP7, coordinated by the Pascale Institute and the focus of this study protocol, is responsible for developing a national platform for the multi-omic profiling of cancer patients eligible for precision medicine treatments, with the goal of supporting clinical decision-making.

DETAILED DESCRIPTION:
The study is multicentric, observational, non-interventional, and both prospective and retrospective.

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate in the study
* Age >18 years
* Performance status (PS) 0-1
* Availability of biological samples for multi-omic profiling
* Availability of radiological images for radiomic assessments
* Patients with metastatic disease, i.e., stage IV (except for melanoma, where stage II/III patients eligible for adjuvant therapy may also be considered)
* Patients eligible for targeted therapy and/or immunotherapy
* Patients with aggressive neoplasms, including melanoma, non-small cell lung carcinoma (NSCLC), colon carcinoma (BRAF-mutated, MSI), triple-negative breast cancer, ovarian cancer, and cholangiocarcinoma.

Exclusion Criteria:

* Previous line of immunotherapy or targeted therapy
* Previous radiotherapy at the sites of the most recent diagnostic biopsy
* Most recent diagnostic biopsy performed >24 months before enrollment
* Absence of measurable lesions
* Presence of active or untreated brain metastases or leptomeningeal carcinomatosis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oncologic patients eligible for targeted therapy and/or immunotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Disease progression | approximately 3 years
  Rate of metastatic patients with disease progression (PD) within 3 months from the start of targeted therapy and/or immunotherapy, or disease recurrence rate at 6 months in patients undergoing adjuvant therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Antonella De Luca, Principal Investigator — IRCCS I.N.T. "G. Pascale"
Locations (1):
- Istituto Nazionale Tumori di Napoli - IRCCS - Fondazione G. Pascale, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No